CLINICAL TRIAL: NCT00999297
Title: Effect of 4-week Dihydrocapsiate Ingestion on Resting Metabolic Rate: A Double-blind Randomized Parallel Arm Study
Brief Title: Effect of 4-week Dihydrocapsiate Ingestion on Resting Metabolic Rate
Acronym: CAPSPAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Ajinomoto USA, INC. (Industry)
Responsible Party: Principal Investigator, Eric Ravussin, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBRC 28016; PBRC28016 (Other: Ajinomoto Co., Inc)
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Weight
Keywords: thermogenesis; respiratory quotient; fat oxidation
MeSH Terms: conditions — Obesity; Body Weight | interventions — capsiate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sugar pill (Placebo o mg/d) (Placebo Comparator): 0 mg/d sugar pill
  Interventions: Other: Dihydrocapsiate
- Dihydrocapsiate (Active Comparator): Drug 3 mg/d or 9 mg/d including Placebo
  Interventions: Other: Dihydrocapsiate
- 3 mg/d or 9 mg/d Dihydrocapsiate (Active Comparator): Drug including Placebo
  Interventions: Other: Dihydrocapsiate

INTERVENTIONS:
Other: Dihydrocapsiate — Capsules will contain dihydrocapsiate 3 mg/d or 9 mg/d or placebo
  Other Names: Natural Substances present in chili pepper
  Arms: Sugar pill (Placebo o mg/d)
Other: Dihydrocapsiate — Capsules will contain dihydrocapsiate 3 mg/d or 9 mg/d or placebo
  Other Names: Natural Substances present in chili pepper
  Arms: Dihydrocapsiate
Other: Dihydrocapsiate — Capsules will contain dihydrocapsiate 3 mg/d or 9 mg/d or placebo
  Other Names: Natural Substances present in chili pepper
  Arms: 3 mg/d or 9 mg/d Dihydrocapsiate

SUMMARY:
A 4 week intake of drug to find a natural substance that may modify energy balance and may enhance health in combination with lifestyle changes with possible decrease in body weight.

DETAILED DESCRIPTION:
This study is a double-blind, placebo-controlled, single center, randomized, parallel arm clinical trial to test the impact of Dihydrocapsiate (placebo, 3 and 9 mg/d) ingested for 4 weeks on resting metabolic rate and fat oxidation measured by indirect calorimetry.

ELIGIBILITY:
Inclusion Criteria:

* Men between 20-60 years old
* Healthy as assessed by medical history and standard medical exam
* Weight-stable
* Body mass index of 25 to 34.9 kg/m2
* Non-smoker
* Sedentary lifestyle: not being physically active grater than 3 days/week for 20 min each time for the previous 6 months, and not participating in regular resistance exercise.

Exclusion Criteria:

* Subjects enrolled in a diet to increase or decrease body weight
* Special diet or food aversiions to common foods
* Has allergy to chilli pepper
* Eating chilli peppers on a daily basis
* Usually consuming more than 2 cups of tea or coffee/day
* Usually consuming more than 4 cans of caffeinated soft drinks a day
* Usually consuming more than 3 standard alcohol drinks/day
* Regular use of medications (weight loss drugs, drugs affecting energy metabolism, drugs for depression)
* Usual intake of illicit substances
* Claustrophobia
* Participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The consumption of dihydrocapsiate will significantly increase resting energy expenditure and fat oxidation | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Result] Galgani JE, Ryan DH, Ravussin E. Effect of capsinoids on energy metabolism in human subjects. Br J Nutr. 2010 Jan;103(1):38-42. doi: 10.1017/S0007114509991358. Epub 2009 Aug 12. PMID 19671203
- [Derived] Galgani JE, Ravussin E. Effect of dihydrocapsiate on resting metabolic rate in humans. Am J Clin Nutr. 2010 Nov;92(5):1089-93. doi: 10.3945/ajcn.2010.30036. Epub 2010 Sep 8. PMID 20826626
- See also: Effect of capsinoids on energy metabolism in human subjects — http://journals.cambridge.org/download.php?file=%2FBJN%2FBJN103_01%2FS0007114509991358a.pdf&code=1af15165e3c2df5c00062d1042e9273c